CLINICAL TRIAL: NCT05820529
Title: Effect of Adenotonsillectomy on Velopharyngeal Valve Mechanism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Mohamed Abdallah, Doctor, Assiut University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Effect of AT on VPV
Record Dates: First submitted 2023-03-20; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Velopharyngeal Insufficiency
MeSH Terms: conditions — Velopharyngeal Insufficiency | interventions — Adenoidectomy; Tonsillectomy

STUDY DESIGN:
Intervention Model Description: We will do Adenotonsillectomy by three different technique
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Effect of Adenotonsillectomy in velopharyngeal valve mechanism (Other): We do adenotonsillectomy and show its effect in velopharyngeal valve
  Interventions: Procedure: adenotonsillectomy; Procedure: adenoidectomy; Procedure: tonsillectomy
- Effect of Adenoidectomy in velopharyngeal valve mechanism (Other): We do adenoidectomy and show its effect in velopharyngeal valve
  Interventions: Procedure: adenoidectomy
- Effect of tonsillectomy in velopharyngeal valve mechanism (Other): We do tonsillectomy and show its effect in velopharyngeal valve
  Interventions: Procedure: tonsillectomy

INTERVENTIONS:
Procedure: adenotonsillectomy — removal of adenoid,tonsil in one session
  Arms: Effect of Adenotonsillectomy in velopharyngeal valve mechanism
Procedure: adenoidectomy — removal of adenoid
  Arms: Effect of Adenoidectomy in velopharyngeal valve mechanism; Effect of Adenotonsillectomy in velopharyngeal valve mechanism
Procedure: tonsillectomy — removal of tonsil
  Arms: Effect of Adenotonsillectomy in velopharyngeal valve mechanism; Effect of tonsillectomy in velopharyngeal valve mechanism

SUMMARY:
1. To assess safety of tonsillectomy, adenoidectomy or adenotonsillectomy result toVelopharyngeal Valve Mechanism.
2. To predict and prevent post adenotonsillectomy velopharyngeal dysfunction.

DETAILED DESCRIPTION:
INTRODUCTION The velopharyngeal mechanism consists of a muscular valve that extends from the posterior surface of the hard palate to the posterior pharyngeal wall and includes the velum, lateral pharyngeal walls and the posterior pharyngeal wall .The function of the velopharyngeal mechanism is to create a tight seal between the velum and pharyngeal walls to separate the oral and nasal cavities for various purposes, including speech. Velopharyngeal closure is accomplished through the contraction of several velopharyngeal muscles including the levator veli palatini, musculus uvulae, superior pharyngeal constrictor, palatopharyngeus, palatoglossus, and salpingopharyngeus. The tensor veli palatini is thought to be responsible for eustachian tube function.(1) Velopharyngeal closure patterns may be classified as follows: coronal, where there is predominant soft palate movement toward the posterior pharyngeal wall; sagittal, where there is predominant movement of the lateral pharyngeal walls toward the pharynx midline, circular, where balanced movements of lateral pharyngeal walls and soft palate are observed; circular with Passavant's ridge, where the circular closure is associated with the development of a mucosal fold named Passavant's ridge on the posterior pharyngeal wall.

Velopharyngeal dysfunction (VPD) is a condition where the velopharyngeal valve does not close consistently and completely during the production of oral sounds. Velopharyngeal dysfunction can be caused by abnormal anatomy (velopharyngeal insufficiency), abnormal neurophysiology (velopharyngeal incompetence),or particular articulation errors (velopharyngeal mislearning)(2). Velopharyngeal dysfunction (VPD) is a generic term which describes a set of disorders resulting in the 3 leakage of air into the nasal passages during speech production. As a result, speech samples can demonstrate hypernasality, nasal emissions, and poor intelligibility.(3) Aetiologies of velopharyngeal insufficiency:( Occult submucous cleft palate, Neuromuscular disorder, Residual adenoid tissue, Classical submucous cleft palate, Poor palatal mobility, Behavioural disorder, Normal palate, 22q11 deletion, Postoperative nasopharyngitis, Scarring from tonsillectomy ).(4) Hypertrophic tonsils can be so large that they push against the posterior faucial pillars and intrude into the pharynx. This can easily be seen through nasopharyngoscopy. When this occurs, it can cause both a functional and mechanical interference with lateral pharyngeal wall movement. In rare cases, a tonsil (or both) is so large that it extends up to the area between the velum and posterior pharyngeal wall, thus interfering with velopharyngeal closure. When hypertrophic tonsils interfere with velopharyngeal function (and also affect the airway(5), this can be corrected with a tonsillectomy. Most children actually have veloadenoidal closure because the adenoids are in the place of normal velar contact. Adenoid tissue is most prominent in very young children but begins to slowly atrophy around the age of 6. With the onset of puberty, there can be significant, and sometimes sudden, atrophy of the adenoid tissue, causing an increase in the distance between the velum and posterior pharyngeal wall. If the velum is normal, it stretches to accommodate the difference in the depth of the pharynx; thus, normal velopharyngeal closure is maintained(6). 15 non-cleft palate children who developed velopharyngeal incompetence (VPI) after adenotonsillectomy. Eight boys and 7 girls with a mean age of 6.2 years (range 4.3-11 years) were treated between 1970 and 1993. After 2 years conservative management to allow for spontaneous resolution, only (7 children) 47% achieved normal resonance. Speech therapy was employed mainly for those 4 patients with unrelated articulation errors. Fifty-three percent (8 children) required surgery for persistent hypernasality and in 6 a pharyngoplasty was performed and in one child a posterior pharyngeal cartilage graft was inserted. One case is still to have surgical intervention. Half of the non-cleft children who develop VPI after adenotonsillectomy will respond to conservative management.(7) Retrospective data collection was performed for patients seen in the Great Ormond Street Hospital for Children multidisciplinary VPI clinic from the 1st of January 2015 until 30th of April 2020. Paediatric patients with previous adenotonsillar surgery and no evidence of cleft palate or speech and language disorder were included in the study.29patients met the inclusion criteria, with 16 having previous adenotonsillectomy and 13 isolated adenoidectomy.Severe hypernasality was noted in 3 patients, while in 20 cases moderate or mild hypernasality was found. There were no patients with normal speech. Ten patients were treated with speech therapy alone, whereas surgical intervention was required in seventeen cases. In the population who received treatment and had adequately recorded follow-up, improvement in speech was noted in 86.9%, with 30.4% having oral resonance on last review. Of the patients with severe hypernasality, all improved but had some persistent hyper nasality on last clinic review(8).

ELIGIBILITY:
Inclusion Criteria:

Children patients (aged from 4yrs to 12yrs) who will be undergone adenoidectomy or tonsillectomy or adenotonsillectomy

Exclusion Criteria:

* Clinical diagnosis of cleft palate.
* Clinical diagnosis of submucous cleft palate
* Neuromuscular disorders.
* Patients with craniofacial syndromes.
* Patient with mental retardation

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of post adenotonsillectomy velopharyngeal dysfunction. | one year
  Velopharyngeal dysfunction will be assessed by doing Fiberooptic endoscopic evaluation preoperative and postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Azzam Abdel-Razek, Professor, Principal Investigator — Assiut University ENT Department; Mahmoud Aly Ragae, Lecturer, Study Director — Assiut University ENT Department; Hanan Abd El Rashed Mohamed, Lecturer, Study Director — Assiut University ENT Department
Locations (1):
- ENT Department, Asyut, Egypt

REFERENCES:
- [Background] Perry JL. Anatomy and physiology of the velopharyngeal mechanism. Semin Speech Lang. 2011 May;32(2):83-92. doi: 10.1055/s-0031-1277712. Epub 2011 Sep 26. PMID 21948636
- [Background] Kummer AW. Types and causes of velopharyngeal dysfunction. Semin Speech Lang. 2011 May;32(2):150-8. doi: 10.1055/s-0031-1277717. Epub 2011 Sep 26. PMID 21948641
- [Background] Lewis JR, Andreassen ML, Leeper HA, Macrae DL, Thomas J. Vocal characteristics of children with cleft lip/palate and associated velopharyngeal incompetence. J Otolaryngol. 1993 Apr;22(2):113-7. PMID 8515508
- [Background] Saunders NC, Hartley BE, Sell D, Sommerlad B. Velopharyngeal insufficiency following adenoidectomy. Clin Otolaryngol Allied Sci. 2004 Dec;29(6):686-8. doi: 10.1111/j.1365-2273.2004.00870.x. PMID 15533160
- [Background] Finkelstein Y, Zohar Y, Nachmani A, Talmi YP, Lerner MA, Hauben DJ, Frydman M. The otolaryngologist and the patient with velocardiofacial syndrome. Arch Otolaryngol Head Neck Surg. 1993 May;119(5):563-9. doi: 10.1001/archotol.1993.01880170089019. PMID 8484947
- [Background] Siegel-Sadewitz VL, Shprintzen RJ. Changes in velopharyngeal valving with age. Int J Pediatr Otorhinolaryngol. 1986 Apr;11(2):171-82. doi: 10.1016/s0165-5876(86)80011-8. PMID 3744698
- [Background] Ng SK, Lee DL, Li AM, Wing YK, Tong MC. Reproducibility of clinical grading of tonsillar size. Arch Otolaryngol Head Neck Surg. 2010 Feb;136(2):159-62. doi: 10.1001/archoto.2009.170. PMID 20157062